CLINICAL TRIAL: NCT06443073
Title: The Mere-measurement Effect in Patient-reported Outcomes: A Randomized Control Trial With Speech Pathology Patients
Brief Title: The Mere-measurement Effect of Patient-reported Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Preston Long, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ECS 2153/2023
Record Dates: First submitted 2024-04-15; First posted 2024-06-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Measurement, Psychological Stress; Speech Disorders; Assessment, Self
MeSH Terms: conditions — Stress, Psychological; Speech Disorders | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control: unhealthy (No Intervention): Participants with a speech disorder who do not receive the intervention and only complete the outcomes.
- Control: healthy (No Intervention): Participants without a speech disorder who do not receive the intervention and only complete the outcomes.
- Experimental groups (Experimental): Four groups receiving different rates of questionnaire exposure and wording at either two or four week intervals.
  Interventions: Other: Patient-reported outcomes for speech disorders: positive

INTERVENTIONS:
Other: Patient-reported outcomes for speech disorders: positive — The Communicative Participation Item Bank (CPIB) aims to assess communication participation in all kinds of communication disorders. The Voice Self-Efficacy Questionnaire (VSEQ) monitors self-efficacy in individuals with self-declared voice problems before and after interventions. The Vocal Fatigue Handicap Questionnaire (VFHQ) and the Vocal Fatigue Index (VFI) aim at reflecting vocal fatigue. Both have been adapted to reflect purely positive wording.
  Other Names: Patient-reported outcomes for speech disorders: negative
  Arms: Experimental groups

SUMMARY:
The use of patient-reported outcome (PROs) have become increasingly commonplace across many healthcare settings over the past two decades. The value of PROs is now acknowledged by healthcare providers and patients alike. However, to date, little is known about the best practices for formulating PRO measures (PROMS), but even more specifically, the effect had on the responding patients as a result of item word choice, emotional valence, or frequency of use. That is, 1) does the positive or negative wording of items affect the patient's perspective on the latent variable, 2) is there a degree of subliminal influence or measurement effects on their behaviour resulting from exposure to PROs, and finally, 3) is such an effect amplified with repeated exposure?

DETAILED DESCRIPTION:
There is currently sufficient evidence to suggest that attributes such as the wording of questions, their presentation order, the context where they are asked, and the item's social sensitivity (e.g. I do not abuse my prescriptions), have an effect on participant responses (1,2). This family of variables are most oft referred to as method effects. Method effects largely regard the phenomenon in which the presentation of an item affects the participant's response independent of the content in question. The end goal within this area of study is to correct for any response bias resulting from the items used. This research primarily concerns psychometrics. It is important to note that while method effects relate to the research questions proposed, it is not the key feature of interest. The ensuing inquiry will not simply focus directly on changes to item responses, but instead, on changes to patient perceptions and behaviours as a result of their exposure to the measures themselves. This has been coined the mere-measurement effect (3) Research supports the claim that asking certain questions can influence behaviours on the same topic (4,5). For example, a randomized-control trial was conducted to assess the impact of asking questions pertaining to blood donation habits of the participants. The researchers found that the subjects whom were asked about their habits were significantly more likely to donate blood than their control counter parts at the following blood-drive (6). Other researchers found that when clinicians did not ask patients with Attention Deficit Hyperactivity Disorder (ADHD) to report whether they were currently medicated on a disease-related severity questionnaire, patients were more likely to report un-medicated symptomologies (7). In other words, patients on ADHD medications responded more symptomatically similar to their un-medicated selves when their medication status was not included on the questionnaire. This suggests that the medication status item itself, may have mitigated ADHD symptoms by bringing the patient's treatment into a higher state of awareness/directing attention.

Thus, it may be that asking patients about their intent to have an operation increases the likelihood of them opting for it, or, that asking them about their exercise increases their physical activity level. If so, this may have significant implications for the effect of routinely collecting patient-reported outcomes (PROs), as well as for utilizing measurements as interventions. However, before value can be attached to such an effect, first the presence and strength must be evaluated in the patient-specific context.

To date, no mere-measurement effect factors have been investigated in the context of patient-reported outcomes measures (PROMs) and particularly not in regard to how they may influence patient perceptions and behaviours. Therefore, exploration of this family of effects must be reduced to a few key anticipated features, namely, emotional valence (positive/negative) and frequency. For instance, would wording a cleft-lip question negatively, such as "I do not like my face", actually decrease the patient's preference for their own face, and, does repeated exposure to this question increase the magnitude of the effect.

This randomized controlled trial (RCT) review will be the first to the authors' knowledge to examine if measuring patient- reported outcomes directly effects their corresponding behaviour, and if this effect can be attributed in part to item wording and/or frequency of exposure.

PROMs & Speech Disorders Three recent reviews regarding patient-reported outcomes in speech pathologies were identified (8,9,10). Francis et al. list a number of PRO measures that were designed for administration with subjects with any kind of voice disorders. The Evaluating Voice Disability-Quality of Life Questionaire (EVD-QOL) aims at assessing the general range of functional problems in voice disorders. The 30-items Voice Handicap Index (VHI) and its 10-items short version VHI-10 aim at providing a psychometrically robust voice diasability/handicap inventory. The Voice-Related Quality of Life (V-RQOL) aims at measuring the impact of voice problems on the quality of life. The Voice Activity and Participation Profile (VAPP) aims at identifying voice activity limitation and participation restriction separately. The Voice Symptom Scale (VoiSS) is an inventory of voice symptoms for assessing baseline pathology and response to change. The Communicative Participation Item Bank (CPIB) aims at assessing communication participation in all kinds of communication disorders. The Voice Self-Efficacy Questionnaire (VSEQ) monitors self-efficacy in individuals with self-declared voice problems before and after interventions. The Vocal Fatigue Handicap Questionnaire (VFHQ) and the Vocal Fatigue Index (VFI) aim at reflecting vocal fatigue.

Additional PROs include the Aging Voice Index, the Evaluation of the Ability to Sing Easily, the Glottal Function Index, the Linear Analog Scale of Assessment of Voice Quality, the Speech Disability Questionnaire, the Trans Woman Voice Questionnaire, the Vocal Cord Dysfunction Questionnaire, and the Vocal Tract Discomfort Scale Slavych, Zraick & Ruleman, 2021.

The researchers have opted to use the CPIB and the VHI because these are well established and the former covers all kinds of communication disorders, while the VHI is using particularly negative wording in its original form.

1.2 STUDY RATIONALE The purpose of the mere-measurement study is to identify the most advantageous way to measure outcomes for patients. This will be accomplished by collecting measures on the same topic at different time intervals and with different wording of questions. The findings of this study should help researchers and clinicians collect measurements from patients in the least burdensome and most beneficial manner possible.

The primary objective of the mere-measurement study is to assess the effects of different collection methods on the responders wellbeing.

The secondary objectives of this study are to:

* What frequency of collection is best for patients?
* What style of question wording is best for patients?

Research Questions:

* Does the assigned positivity or negativity of an item effect patient perception or behaviour on the topic inquired?
* Does frequency of exposure to an item have an effect on patient perception or behaviour of the topic inquired?

Hypotheses:

H1 = The more a patient reads and responds to questions about their speech condition the more their speech condition will be affected.

H2 = The directionality of impact on a speech condition will be congruent with the emotional valence of the items used.

STUDY DESIGN Once a subject has agreed to participate in this study, they will be asked to complete online questionnaires as well as record their voice reading a collection of random words 2-4 times.

This study follows a 2x2 design. Participants will be randomly assigned to one of four groups. Randomization will be accomplished by using the MUW randomizer. Participants will be stratified by education and speech disorder type. The healthy case control group will undergo case matching to ensure comparability across groups. Each group will receive two brief speech pathology severity questionnaires but at different frequencies, and with slight adjustments to the wording. Depending on the experimental group, a subject will complete the questionnaires either two or four times, separated each time by one week. The questionnaires, in all groups, will take approximately 15 minutes to complete. Lastly, at the very start and once at the very end of the study, every participant will also be asked to record a brief 45 second audio file in the online survey as well as complete two additional psychological questionnaires.

The measures in this study cover the following tools (complete measures are uploaded in the ECS):

* A patient-reported outcome on voice health - Voice Handicap Index (VHI) or Voice Handicap Index Positively adapted (VHI-PA)
* A patient-reported outcome on speech health - Communicative Participation Item Bank (CPIB) or Communicative Participation Item Bank Positively adapted (CPIB-PA)
* A self-esteem stability scale - Self-Esteem Stability Scale (SESS)
* A self-esteem scale - Rosenberg Self-Esteem Scale (RSS)
* Two question measure of disease impact (2DB)
* A single-question measure of disease activity (1DS)
* Audio recording of text read aloud (ARec)

Study population All patients with Muscle tension dysphonia, Inducible laryngeal obstruction, Amyotrophic lateral sclerosis (ALS), suffering from a stroke or other brain injury/damage/trauma, (aphasia, dysarthria), and Parkinson's disease will be targeted for recruitment. There are no geographic location requirements. The participation schedule can be found below. Patients will be informed of the schedule in advance. A subject must complete any respective sampling epoch within 48 hours of the prescribed date in order to qualify as completed. Subjects must also have strong English skills and be technologically savvy to participate. Only adults will be included in the study.

Study Design Flow Group 1: High frequency-negative: 1 week between each collection

1. Demographics, VHI, CPIB, SESS, RSS, 1DS, 1DB, ARec*
2. VHI, CPIB, SE, SSE, 1DS, 2DB, ARec
3. VHI, CPIB, SE, SSE, 1DS, 2DB, ARec
4. VHI, CPIB, SE, SSE, 1DS, 2DB, ARec Group 2: High frequency-positive: 1 week between each collection

<!-- -->

1. Demographics, VHI-PA, CPIB-PA, SESS, RSS, 1DS, 2DB, ARec*
2. VHI-PA, CPIB-PA, SE, SSE, 1DS, 2DB, ARec
3. VHI-PA, CPIB-PA, SE, SSE, 1DS, 2DB, ARec
4. VHI-PA, CPIB-PA, SE, SSE, 1DS, 2DB, ARec Group 3: Low frequency-negative: 2 weeks between each collection

1: Demographics, VHI, CPIB, SESS, RSS, 1DS, 2DB, ARec* 2: VHI, CPIB, SE, SSE, 1DS, 2DB, ARec Group 4: Low frequency-positive: 2 weeks between each collection

1. Demographics, VHI-PA, CPIB-PA, SESS, RSS, 1DS, 2DB, 1ARec*
2. VHI-PA, CPIB-PA, SE, SSE, 1DS, 2DB, 1ARec Control: (once at start, once at low frequency completion/final outcome collection, once at high frequency completion)

1: Demographics, ARec x 3

Healthy Control: (once at start, once at low frequency completion/ final outcome collection, once at high frequency completion)

1. Demographics, ARec x 3

   *completed prior to assessments

   *English was chosen as the study language as a wider range of validated assessments exist in this language. The AI used for speech analysis is also best suited for and trained (66%) on English. Lastly, English is the most prolific language (native + secondary speakers) in the world which will facilitate the speed of recruitment.

   Subjects who meet any of the following criteria will be excluded from study entry:

   • Under the age of 18

   NUMBER OF SUBJECTS PARTICIPATING IN THE STUDY Subjects will be randomly separated into six groups including control and healthy control, with approximately 33 subjects per group. A formal power analysis was performed using G*power with parameters sourced from relevant seminal research (Conner et al., 2011; Godin et al., 2011). The following parameters were used for the sample size analysis: two-tailed directionality; effect size of 0.30; a priori computation, anticipated power of 0.95, and an error rate of 0.0023. Means difference tests between independent groups within the t-test family were utilized.

   RECRUITMENT PROCEDURE Recruitment into the mere-measurement study will be performed supported by Probando. Probando is a previously approved patient recruitment service that specializes in online advertising. All recruitment materials are uploaded to the ECS. A description of the Probando recruitment service and procedures can be found as an attachment, as well as the recruitment materials for all subjects including healthy controls and a screenshot of the currently inactive landing page. As a part of their service, Probando uses the study inclusion and exclusion criteria to screen potential interested subjects. If they qualify and permit contact, their contact information will be provided to the MUW researchers for direct outreach. Therefore, all study timings, measures, and data will be distributed and collected only by the study researchers. Patients will be able to withdraw from the study at any time without providing a reason. To limit potential bias, an initial self-report of an official diagnosis is required to participate. Additionally, the patients will also confirm their diagnosis with a checkbox, for the purpose of minimizing the risk of malingering patients. If an individual is highly motivated to participate and does not suffer from a qualifying speech disorder they can still apply to participate as a healthy control. Furthermore, this sample would be more representative of a telemedicine community.

   DATA SOURCES

   Participants' and study data will be recorded in the study database. Study data will be collected at defined time points (see Section 1.5) using a single online format:

   • SoSci survey (www.soscisurvey.de) is a routinely used, safe, online questionnaire distribution and data retrieval platform. Within this platform, five links will be created, one for each group. These will connect subjects to the questionnaires and to the instructions for capturing the audio file.

   An email address for every participant will be required for communication and dissemination of participation credits. All individuals with access to participants' personal information are obligated to respect their privacy and only use and disclose their information as described in the informed consent document.

   Demographic information and mere-measurement study results are secured against unauthorized access. Security measures reduce the risk of unauthorized individuals accessing subject personal information, but such risks cannot be entirely eliminated. All audio recordings will be stored only for the duration of the study. Upon closure, they will be deleted.

   The information collected from the mere-measurement study will be kept confidential. Subject personal information will be stored safely at MUW and pseudonymized as discussed in the previous section.

   DATA COLLECTION

   Online, subjects will complete a battery of questionnaires totalling approximately 15-20 minutes of time following the informed consent. Informed consent will be collected online via the SoSci survey tool. The following parameters will be applied to the virtual informed consent:

   • The patient information including the data protection section is displayed above the checkbox. The patients are informed about what happens to their data, their benefits, and risks in sufficient detail but simple detail in this section.

   • The checkbox says that patients have read and understood the text and that they agree.

   • The patients will confirm their diagnosis with a checkbox, for the purpose of minimizing the risk of malingering patients Depending on the group assigned, a participant will have to complete this battery either 2 or 4 times. The control and healthy group will complete only demographics questions and the audio recordings, no PROMs will be collected. The four intervention groups will be randomized using a digital randomization tool provided by the MUW (https://www.meduniwien.ac.at/randomizer/ ).

   All patients, across all intervention groups, will complete the read-aloud activity prior to the first collection of PROMs. This will serve as the baseline for later comparison. Following the first recording, all subsequent recordings will be completed after completing the PROMs. An electronic bank transfer form (MUW standard bank form) will be emailed to participants at the end of the study to complete the 50€ transfer. These electronic records will be immediately destroyed upon successful completion.

   DATA MANAGEMENT Patient-reported data will be captured using SoSci survey with an account owned by the Center for Outcomes Research. These data will not be transferred outside of the MUW. Data transfers between the investigators of this study will be managed using procedures described in a jointly developed Data Transfer Plan. All data transferred between the two MUW centers, speech pathology and outcome research, will be identified only by a subject ID code, unless otherwise consented by patients and agreed upon in the Data Transfer Plan.

   DATA QUALITY ASSURANCE Patients will consent that pseudonymized patient data will be hosted and analysed at the MUW. MUW will not share the data with any third parties or collaborators. MUW regularly processes medical data and is subject to the GDPR requirements. MUW is responsible for data quality and will perform oversight of the data management of this study. Investigators and study coordinators will receive an initial training session on the protocol, study flow, study database, survey tool, documentation, and expectations, and any applicable study processes. Access to data for secondary use cases will not be enabled.

   SOURCE DATA DOCUMENTATION

   Source documents (electronic) are those in which participant data are recorded and documented for the first time. The source documentation for this study will be:
   * Participant demographic information and eligibility assessment
   * Completed Informed Consent Forms
   * Audio recordings
   * Completed PROMs

ELIGIBILITY:
Inclusion Criteria:

All patients will be required to have a qualifying disorder known to effect speech as identified below. Patients who meet the eligibility criteria will be invited to participate in the study by the researchers. Eligibility will be assessed prior to enrolment recruitment screening. AKH patients are not targeted for this study. All patients, regardless of geographic location around the world, can be recruited. The study is entirely online.

Subjects must meet the following inclusion criteria for study entry:

* Strong English skills*
* Technology savvy - able to complete online questionnaire
* Suffering from one of the following:

  * Muscle tension dysphonia
  * Inducible laryngeal obstruction
  * Amyotrophic lateral sclerosis (ALS)
  * Patients after a stroke or other brain injury/damage/trauma, (aphasia, dysarthria)
  * Parkinson's disease

Exclusion Criteria:

* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
audio recording of a standardized text | Baseline and at each experimental instance occuring once a week for up to four weeks
  • An audio recording of a standardized text, with the order of the paragraphs randomized in between every exposure. This text was adapted from the standard "Rainbow Passage" read aloud assessment with the field of speech pathologies (Dietsch et al., 2023). Artificial intelligence - ChatGPT - was used to recreate novel text of the same length and difficulty as the "Rainbow Passage" which is called "In the heart of a lush valley" (the text is uploaded in the ECS). An adapted version was opted for to eliminate the possibility of previous exposure.

SECONDARY OUTCOMES:
Self-Esteem Stability Scale (SESS) | Baseline and at each experimental instance occuring once a week for up to four weeks
  A three-item self-esteem stability scale - Self-Esteem Stability Scale (SESS). Scores range from 1-6 with higher scores suggesting less stability.
Disease activity (1DS) | Baseline and at each experimental instance occuring once a week for up to four weeks
  A single-question measure of disease activity (1DS). Score range of 1-5 with higher scores denoting more activity.
A self-esteem scale - Rosenberg Self-Esteem Scale (RSS) | Baseline and at each experimental instance occuring once a week for up to four weeks
  A nine-item scale measuring self-esteem. Score range of 1-4 with high scores denoting lower self-esteem.
Disease Impact | Baseline and at each experimental instance occuring once a week for up to four weeks
  Two-question measure of disease impact (2DB). Score range of 1-4 with higher scores denoting more impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Preston Long, Vienna, Austria

REFERENCES:
- [Background] Schwarz, N. (1999). Self-reports: How the questions shape the answers. American Psychologist, 54(2), 93-105. https://doi.org/10.1037/0003-066X.54.2.93
- [Background] Näher, A.-F., & Krumpal, I. (2012). Asking sensitive questions: The impact of forgiving wording and question context on social desirability bias. Quality & Quantity: International Journal of Methodology, 46(5), 1601-1616. https://doi.org/10.1007/s11135-011-9469-2
- [Background] Morwitz, V. G., Johnson, E., & Schmittlein, D. (1993). Does measuring intent change behavior?. Journal of consumer research, 20(1), 46-61.
- [Background] Sandberg T, Conner M. A mere measurement effect for anticipated regret: impacts on cervical screening attendance. Br J Soc Psychol. 2009 Jun;48(Pt 2):221-36. doi: 10.1348/014466608X347001. Epub 2008 Sep 12. PMID 18793492
- [Background] Godin G, Sheeran P, Conner M, Delage G, Germain M, Belanger-Gravel A, Naccache H. Which survey questions change behavior? Randomized controlled trial of mere measurement interventions. Health Psychol. 2010 Nov;29(6):636-44. doi: 10.1037/a0021131. PMID 20939639
- [Background] Godin G, Sheeran P, Conner M, Germain M. Asking questions changes behavior: mere measurement effects on frequency of blood donation. Health Psychol. 2008 Mar;27(2):179-84. doi: 10.1037/0278-6133.27.2.179. PMID 18377136
- [Background] Lineweaver TT, Kercood S, Gabor AJ, Cervantes J, Laine A, Baker E. The effect of medication and question wording on self-reported symptoms and their accuracy in young adults with attention-deficit/hyperactivity disorder. Br J Clin Psychol. 2021 Jun;60(2):252-269. doi: 10.1111/bjc.12276. Epub 2021 Jan 4. PMID 33393098
- [Background] Cohen ML, Hula WD. Patient-Reported Outcomes and Evidence-Based Practice in Speech-Language Pathology. Am J Speech Lang Pathol. 2020 Feb 7;29(1):357-370. doi: 10.1044/2019_AJSLP-19-00076. Epub 2020 Feb 3. PMID 32011905
- [Background] Francis DO, Daniero JJ, Hovis KL, Sathe N, Jacobson B, Penson DF, Feurer ID, McPheeters ML. Voice-Related Patient-Reported Outcome Measures: A Systematic Review of Instrument Development and Validation. J Speech Lang Hear Res. 2017 Jan 1;60(1):62-88. doi: 10.1044/2016_JSLHR-S-16-0022. PMID 28030869
- [Background] Slavych BK, Zraick RI, Ruleman A. A Systematic Review of Voice-Related Patient-Reported Outcome Measures for Use with Adults. J Voice. 2024 Mar;38(2):544.e1-544.e14. doi: 10.1016/j.jvoice.2021.09.032. Epub 2021 Nov 12. PMID 34782227

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT06443073/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT06443073/ICF_001.pdf